CLINICAL TRIAL: NCT00787930
Title: Bipolar Disorder in Late Life (Evaluation of MRI Hyperintensities and DTI in Bipolar Disorder)
Brief Title: Bipolar Disorder in Late Life
Acronym: BPD
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00007867
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Bipolar Disorder
Keywords: BPD
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA collected for genetic databank.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Manic Subject with DWM Hyperintensities >2: Subjects with acute mania who were treated with naturalistic protocol (starting with valproic acid) who had a BOYKO DWM Hyperintensity rating >2 and a YMRS <15 at week 3.
  Interventions: Drug: Valproic Acid
- Manic Subjects with DWM Hyperintensities <3: Subjects with acute mania who were treated with naturalistic protocol (starting with valproic acid)who had a BOYKO DWM Hyperintensity rating <3 and a YMRS <15 at week 3.
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid — Tablets, 250mg-3000mg
  Other Names: Depakote

SUMMARY:
The purpose of this study is to look at certain structural changes in the brain in people with bipolar disorder or those with a history of Bipolar disorder.

DETAILED DESCRIPTION:
Individuals with bipolar disorder or those with a history of bipolar disorder may have certain structural changes in their brain. The purpose of this study is to look at those changes, as well as the assessment of risk factors for bipolar disorders, involving both social and psychological aspects of behavior, age, education, marital relations, nutrition, physical activity, etc., compared with persons not having bipolar disorder. These changes in the brain will be measured by Magnetic Resonance Imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV diagnosis of bipolar Disorder, Manic and mixed episodes.
2. 18 years of age and older, male or female, any race.
3. Capacity to give informed consent and follow study procedures.

Exclusion Criteria:

1. History of alcohol/drug dependence
2. Any metal or pacemaker in the body which precludes MRI
3. Pregnancy
4. Dementia or other primary psychiatric disorders including substance abuse/dependence, anxiety disorders, schizophrenia
5. For controls, numbers one through four above as well as any history of depression or the use of antidepressants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects recruited from the adult inpatient and outpatient psychiatric clinics at Duke University Medical Center and John Umstead Hospital (Butner, NC).
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2005-10; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L Beyer, M.D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 2005-2009 from the inpatient units and Duke University Medical Center and John Umstead Hospital and the outpatient clinics at DUMC.
Pre-assignment Details: Only subjects currently in a manic episode were recruited for the acute treatment protocol substudy.
Groups:
- Naturalistic Treatment: Acutely manic subjects were treated using the Systematic Treatment Enhancement Program for Bipolar Disorder (STEP-BD) expert consensus guidelines beginning with valproic acid (titrated to therapeutic levels) over a three week period. If there was a non-response to this intervention, then a subject would continue acute treatment using other interventions indicated by STEP-BD protocols. After stabilization, subjects were followed monthly up to a year's duration and treated using the STEP-BD expert consensus guidelines.
Period: Acute Treatment -- 3 Weeks
Arm/Group | Naturalistic Treatment
Started | 19
Completed | 19
Not Completed | 0
Period: Continuation Treatment -- up to 12 Month
Arm/Group | Naturalistic Treatment
Started | 19
Completed | 16
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Naturalistic Treatment
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.68 (17.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Boyko DWM Hyperintensity Value >2 in Subjects Who Received Acute Treatment for Mania
Description: Subject with acute mania were treated for 3 weeks with STEP-BD protocol using valproic acid as the primary intervention. Subject MRI's were evaluated for the presence of deep white matter hyperintensities (DWM) (>2 on the the Boyko Classification). Boyko lesion classification system assesses DWM hyperintensities as follows: 0 = absent, 1 = punctate, 2 = rounded <5 mm, 3 = irregular >5 mm, 4 = confluent lesions.
Time Frame: 3 weeks
Population: All subjects in an acute manic state who were treated with specified protocol.
Measure: Number; unit: participants
Groups:
- Responders to Acute Treatment: Subjects in an acute manic episode who responded to treatment as measured by a Young Mania Rating Scale (YMRS) <15 by week 3, which was the protocol-defined determination point for response to treatment.
- Non-Responders to Acute Treatment: Subjects in an acute manic episode who did not respond to treatment as measured by a YMRS >15 by week 3.
Arm/Group | Responders to Acute Treatment | Non-Responders to Acute Treatment
Number analyzed (Participants) | 10 | 9
participants | 10 | 9
Statistical Analysis 1: Comparison: Responders to Acute Treatment vs Non-Responders to Acute Treatment; Test type: Superiority or Other; p > 0.05, Chi-squared — a priori threshold for significance was 0.05

2. Primary Outcome: Boyko DWM Hyperintensity Value >2 in Subjects Who Received Continuation Treatment
Description: Subject were evaluated for relapse of their mood disorder and for the presence of DWM Hyperintensities (>2 on the the Boyko Classification. Boyko lesion classification system assesses DWM hyperintensities as follows: 0 = absent, 1 = punctate, 2 = rounded <5 mm, 3 = irregular >5 mm, 4 = confluent lesions. Subjects were also assessed for relapse, as defined by the Montgomery-Asberg Depression Rating Scale (MADRS)and the Young Mania Rating Scale (YMRS). Relapse was defined by protocol as either a MADRS scale >15 or a YMRS scale >15.
Time Frame: 12 months
Population: Subjects who completed at least 4-12 months of consistent follow up appointments after stabilization from an acute manic episode. Note that 3 subjects dropped out of continuation treatment.
Measure: Number; unit: participants
Groups:
- Relapse Into Depression or Mania: Subjects who relapsed into a depressive or manic episode within the 12 months following stabilization as measured by the YMRS or MADRS scales.
- Non-relapse Into Depression or Mania: Subjects who had no depressive or manic episodes within the 12 months following stabilization as measured by the YMRS or MADRS scales.
Arm/Group | Relapse Into Depression or Mania | Non-relapse Into Depression or Mania
Number analyzed (Participants) | 9 | 7
participants | 4 | 4
Statistical Analysis 1: Comparison: Relapse Into Depression or Mania vs Non-relapse Into Depression or Mania; Test type: Superiority or Other; p = 1.00, Chi-squared; df=1

3. Secondary Outcome: Boyko Subcortical (SC) Hyperintensity Value >2 in Subjects Who Received Continuation Treatment
Description: Subject were evaluated for relapse of their mood disorder and for the presence of subcortical (SC) Hyperintensities (>2 on the the Boyko Classification). Boyko lesion classification system assesses SC hyperintensities as follows: 0 = absent, 1 = punctate, 2 = rounded <5 mm, 3 = irregular >5 mm, 4 = confluent lesions. Subjects were also assessed for relapse, as defined by the Montgomery-Asberg Depression Rating Scale (MADRS)and the Young Mania Rating Scale (YMRS).
Time Frame: up to 12 months
Population: Number of subjects who who had >2 on the DWM hyperintensity assessment from the Boyko classification system.
Measure: Number; unit: participants
Arm/Group | Relapse Into Depression or Mania | Non-relapse Into Depression or Mania
Number analyzed (Participants) | 9 | 7
participants | 2 | 4
Statistical Analysis 1: Comparison: Relapse Into Depression or Mania vs Non-relapse Into Depression or Mania; Test type: Superiority or Other; p = 0.6056, Chi-squared — No adjustment for multiple comparisons; df=1

4. Secondary Outcome: fa LOFC in Subjects Who Received Continuation Treatment
Description: As an exploratory analysis, subject MRI's were also evaluated using diffusion tensor imaging (DTI) for differences in fractional anisoptery (fa) in the Left Orbitofrontal area (LOFC). FA is a scalar value between zero and one hundred that describes the degree of anisotropy of a diffusion process. A value of zero means that the diffusion is isotropic (unrestricted in all directions). A value of one hundred means that diffusion occurs only along one axis and is fully restricted along all other directions.
Time Frame: up to 12 months
Population: Number of subjects in continuation phase who had MRIs that were able to be processed for DTI data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Relapse Into Depression or Mania: Subjects who relapsed into a depressive or manic episode within the 12 months following stabilization as measured by the Young Mania Rating Scale (YMRS) >15 or Montgomery Asberg Depression Rating Scale (MADRS) scales >15.
  MADRS is an ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients. Scale: 0-60 Higher MADRS scores indicate more severe depression.
  YMRS is an eleven-item, multiple choice diagnostic questionnaire used to measure the severity of manic episodes in patients. Scale: 0-60 Higher YMRS scores indicate more mania.
- Non-relapse Into Depression or Mania: Subjects who had no depressive or manic episodes within the 12 months following stabilization as measured by the Young Mania Rating Scale (YMRS) <15 or Montgomery Asberg Depression Rating Scale (MADRS) scales <15.
  MADRS is an ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients. Scale: 0-60 Higher MADRS scores indicate more severe depression.
  YMRS is an eleven-item, multiple choice diagnostic questionnaire used to measure the severity of manic episodes in patients. Scale: 0-60 Higher YMRS scores indicate more mania.
Arm/Group | Relapse Into Depression or Mania | Non-relapse Into Depression or Mania
Number analyzed (Participants) | 7 | 3
units on a scale | 76.3 (8.18) | 81.4 (1.81)
Statistical Analysis 1: Comparison: Relapse Into Depression or Mania vs Non-relapse Into Depression or Mania; Test type: Non-Inferiority or Equivalence — Exploratory hypothesis; p = 0.081, t-test, 1 sided; missing values: 6 df=7; t-stat estimated value = 1.52, 95% CI 1-sided [lower limit 0], Standard Deviation 8.2

5. Secondary Outcome: fa ROFC in Subjects Who Received Continuation Treatment
Description: As an exploratory analysis, subject MRI's were also evaluated using diffusion tensor imaging (DTI) for differences in fractional anisoptery (fa) in the Right Orbitofrontal area (ROFC). FA is a scalar value between zero and one hundred that describes the degree of anisotropy of a diffusion process. A value of zero means that the diffusion is isotropic (unrestricted in all directions). A value of one hundred means that diffusion occurs only along one axis and is fully restricted along all other directions.
Time Frame: up to 12 months
Population: Number of subjects in continuation phase who had MRIs that were able to be processed for DTI data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Non-relapse Into Depression or Mania: Subjects who relapsed into a depressive or manic episode within the 12 months following stabilization as measured by the Young Mania Rating Scale (YMRS) >15 or Montgomery Asberg Depression Rating Scale (MADRS) scales >15.
  MADRS is an ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients. Scale: 0-60 Higher MADRS scores indicate more severe depression.
  YMRS is an eleven-item, multiple choice diagnostic questionnaire used to measure the severity of manic episodes in patients. Scale: 0-60 Higher YMRS scores indicate more mania.
Arm/Group | Relapse Into Depression or Mania | Non-relapse Into Depression or Mania
Number analyzed (Participants) | 7 | 4
units on a scale | 76.1 (6.56) | 79.8 (1.39)
Statistical Analysis 1: Comparison: Relapse Into Depression or Mania vs Non-relapse Into Depression or Mania; Test type: Non-Inferiority or Equivalence — Exploratory analyses; p = 0.091, t-test, 1 sided — no adjustment for multiple analyses; missing values: 5 df=7; t-stat estimated value = 1.47, 95% CI 1-sided [lower limit 0], Standard Deviation 6.56

ADVERSE EVENTS:
Groups:
- Naturalistic Treatment: Patients were treated acutely using expert consensus guidelines beginning with valproic acid. After stabilization, subjects were followed monthly up to a year's duration and treated using expert consensus guidelines. indicated.
Arm/Group | Naturalistic Treatment
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naturalistic Treatment (N=19)
Lithium Toxicity (Nervous system disorders) | 1 (1) — Patient was readmitted after being found to be lithium toxic. Condition resolved without treatment. No sequela noted.

LIMITATIONS AND CAVEATS:
Acute MRI hypothesis unable to be tested due to high subject response. Five subject scans could not be evaluated by DTI computer program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No